CLINICAL TRIAL: NCT02773862
Title: Prospective Evaluation of the Non-invasive ICP HeadSense Monitor in TBI Patients Undergoing Invasive ICP Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HeadSense Medical (Industry)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-012
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Brain Injuries; Intracranial Hypertension
Keywords: brain injuries; noninvasive monitoring; intracranial pressure
MeSH Terms: conditions — Brain Injuries; Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): ICP monitoring will be done in parallel for both HS-1000 and ICP monitoring via an invasive monitoring device (per clinical protocol without any change in the patient's management). HS-1000 ICP monitoring intervals will last from 30 minutes to 48 hours, continuously depending on the patient's clinical condition.
  Interventions: Device: HS-1000

INTERVENTIONS:
Device: HS-1000

SUMMARY:
Patients with severe traumatic brain injury (TBI) are admitted to the intensive care unit (ICU). Under certain condition (such as a impaired consciousness) the intracranial pressure (ICP) is measured. An increase in the intracranial pressure might suggest secondary neurological deterioration and is considered an alarming symptom. Current practice is to insert an invasive monitor through a burr hole in the skull with the risk of bleeding and infection. Using a new type of ICP monitor (HeadSense) it is possible to measure ICP non-invasively through an acoustic signal.

DETAILED DESCRIPTION:
In this pilot study, the investigators will prospectively collect relevant clinical data on 15 TBI patients with an inserted invasive ICP monitor. Each enrolled patient will be monitored in parallel to the invasive ICP monitor with the HeadSense's ICP monitor. Subjects who meet the study's inclusion and exclusion criteria will be enrolled in the study. Family members will be asked for consent. The patient's clinical condition will be recorded in a case record form (CRF).

Once the patient is inclined with his upper body 30 degrees to the bed and the invasive ICP monitor displays the pressure values, the clinical procedure can begin. Once the HeadSense's monitor is calibrated it is connected to the front end that is placed on the patient's ears. Each recording session will be ½-48 hours long, depending on the patient's clinical condition. In case the ICP monitor is still inserted to the patient's brain in the following day, recording sessions will continue until the ICP monitor is removed.

After the study, the patient's ears will be examined for internal ear infection or irritation that might be caused by the ear buds. Patient adverse events will be documented on the case report forms in case they occurred, and the family or advocate of the patient will be informed. In case of clinical relevant adverse event, appropriate clinical action will be taken.

As the procedure does not affect the patient management, there is no need to provide any specific medical care related to the trial. Patients will receive the relevant clinical care related to their clinical management, without any consideration to their participation in the trial.

Once the data collection is done, results will be analyzed by comparing ICP readings from both devices. The end point of the study is to collect at least half an hour of ICP monitoring for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have an invasive ICP monitoring
* Male or Female in the age range of 18 years and older

Exclusion Criteria:

* Local infection in the ear.
* Pregnant/lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of ICP values obtained by the HS device that correlate to ICP using current standards | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Guus Schoonman, MD, PhD, Principal Investigator — St. Elisabeth/Tweesteden Hospital Tilburg
Locations (1):
- St. Elisabeth Ziekenhuis, Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: No